CLINICAL TRIAL: NCT00442000
Title: Outcomes Comparison of Robotic, Retropubic, and Perineal Prostatectomy
Status: Completed | Type: Observational
Sponsor: Corewell Health East (Other)
Responsible Party: Sponsor
Other Study IDs: E2007-024
Record Dates: First submitted 2007-02-28; First posted 2007-03-01 (Estimated); Last update posted 2012-03-21 (Estimated); Status verified 2012-03

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Prostatectomy

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Prostatectomy — Patients undergoing prostatectomy.

SUMMARY:
Compare peri-operative and postoperative outcomes of the three different surgical approaches to prostatectomy

DETAILED DESCRIPTION:
Existing data collected from Prostatectomy Database study and Urology Database study will be analyzed. Compare peri-operative and postoperative outcomes of the three different surgical approaches to prostatectomy

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* Radical Prostatectomy at William Beaumont Hospital

Exclusion Criteria:

* Dementia

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing prostatectomy at William Beaumont-Royal Oak.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2005-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Feber, M.D., Principal Investigator — Corewell Health East
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States